CLINICAL TRIAL: NCT05363293
Title: A Multiple-dose, Steady-state, Double-blind, Ascending Dose, Safety, Tolerability, Pharmacokinetic Study of AL001 in Patients With Mild to Moderate Alzheimer's Disease and Healthy Adult Subjects ("MAD Study")
Brief Title: Multiple Ascending Dose Safety, Tolerability, PK Study of AL001 in Alzheimer's Disease Patients & Healthy Adult Subjects
Acronym: "MAD"
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alzamend Neuro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL001-ALZ02
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer's Disease; Healthy Non-elderly and Elderly Adults
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Multi-center, placebo-controlled, double-blind, randomized, multiple ascending dose clinical trial to determine the safety and maximum tolerated dose of AL001.
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 1 (Experimental): Participants will be randomized to receive AL001. When adequate safety data are available, a review will be done for all participants to make a dose-escalation or dose and/or regimen modification decision. This will be repeated for each cohort.
  A total of 9 cohorts will receive 5 different dose levels of AL001 in multiple ascending doses under fasted conditions up to tolerability/safety limits.
  Cohort 1 will include 8 AD subjects. In this cohort, 6 active and 2 placebo AD subjects (as per randomization code) will receive the following treatment or placebo:
  • Cohort 1: 60% of 450 mg lithium carbonate equivalent of AL001 (1890 mg AL001 daily ×14 days, given as 3 × 210 mg AL001 capsules TID)
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohorts 2a (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 2a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 2a: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 3a (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 3 will be sub-divided into 2 cohorts: Cohort 3a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 3b (8 AD subjects). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 3a and 3b: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 4a (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 4a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 4a: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 5a (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 5a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 5a: 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohorts 2b (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 2b (8 AD subjects). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 2b: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 3b (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 3b (8 AD subjects). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 3b: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 4b (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 4b (8 AD subjects). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 4b: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  Interventions: Drug: AL001; Other: Placebo
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 5b (Experimental): The data from the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  Cohort 5b (8 AD subjects). Per randomization, there will be 6 active and 2 placebo subjects in each cohort:
  • Cohort 5b: 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID).
  Interventions: Drug: AL001; Other: Placebo

INTERVENTIONS:
Drug: AL001 — a crystal engineered lithium-salicylate-proline lithium delivery product
  Other Names: Alzamend AL001
Other: Placebo — matching placebo formulation

SUMMARY:
This is a Phase 1/2a, multi-center, placebo-controlled, double-blinded, randomized, multiple ascending dose (MAD) clinical trial to determine the safety and maximum tolerated dose of AL001. Up to 72 participants will be randomly assigned to receive study drug (active AL001) or placebo. The study consists of a 4-week screening period, a 14-day treatment period, and a 42-day follow-up period.

DETAILED DESCRIPTION:
This is a Phase 1/2a, multi-center, placebo-controlled, double-blind, randomized, multiple ascending dose (MAD) clinical trial to determine the safety and maximum tolerated dose (MTD) of AL001, a crystal engineered lithium-salicylate-proline lithium delivery product that in nonclinical studies was shown to enhance and prolong the pharmacokinetic (PK) profile of lithium in the brain with enhanced efficacy potential in Alzheimer's models compared to lithium carbonate.

A maximum of approximately 72 participants will be enrolled. Participants will be randomly assigned to receive study drug (active AL001) or placebo in a ratio of 6:2, respectively, with 8 patients in each dosing cohort. Placebos will be pooled and regarded as a comparative cohort for safety.

Cohorts 2a, 3a, 4a and 5a will involve 1:1 healthy non-elderly and elderly subjects; cohorts 1, 2b, 3b, 4b and 5b will involve Alzheimer's subjects. The study will consist of a screening period (Days -28 to -2), a 14-day treatment period, and a 42-day follow-up period.

ELIGIBILITY:
Inclusion Criteria (Alzheimer's Patients):

* Mild to moderate Alzheimer's disease (reasonably good physical health per Investigator's review of medical & surgical history, physical examination incl. neurological examination, 12-lead ECG, vital signs, and clinical laboratory tests)
* Able to understand and provide written informed consent and able to understand and follow instructions during study as determined by Investigator
* Subject and caregiver (if accompanying subject on site) willing to follow study procedures, willing & able to adhere to study restrictions and to be confined at the clinical research center for 16 days
* Fluent in English speaking, reading, and writing (for cognitive testing)
* Availability of medical history to provide information about the cognitive and functional level of the participant and of a qualified source such as the caregiver willing and able to provide information about the cognitive and functional level of the participant
* Males (non-vasectomized and vasectomized) must agree to use barrier contraception during the study until after Study Day 42
* Females must meet criteria if childbearing for contraception or be non-childbearing
* Clinical diagnosis of dementia (neurocognitive disorder) by a qualified clinician based on the DSM-V criteria
* Considered AD Stage 2, 3, or 4 based on the FDA classification
* Mini-Mental State Examination (MMSE) score between 16 and 26, inclusive, at Screening
* Negative result to COVID-19 test at Screening and admission (performed on Day -1)

Exclusion Criteria (Alzheimer's Patients):

* Clinically significant abnormalities (as determined by investigator based on medical history, physical examination, vital sign measurements, ECG findings, or clinical laboratory findings) that may affect subject safety or successful study participation
* Presence or history of any disorder that may prevent the successful completion of the study
* Other severe acute, chronic, or historical medical or psychiatric condition or laboratory abnormality or social circumstance that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in judgment of the Investigator, would make the subject inappropriate for entry into this study
* Evidence of clinically significant hematological, renal, endocrine, pulmonary, cardiovascular, dermatologic, muscular, or allergic disease or disorder (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) that may affect the safety or successful participant of the subject
* Any history or presence of gastrointestinal disease including chronic gastritis, hemorrhagic gastritis, peptic ulcers, duodenitis, diarrhea, or inflammatory bowel disease
* Any presence or history of acute or chronic liver diseases
* Any post-surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the study treatment
* Any history of frequent headache or migraine
* Kidney disease (eGFR <60 mL/minute/1.73 m2)
* Uncontrolled tachy/brady arrhythmias, atrial fibrillation, or coronary heart failure
* Psychiatric or neurological illnesses (other than Alzheimer's disease), e.g., schizophrenia or other psychotic syndromes, Parkinson's disease and related movement disorders, myasthenia gravis, and seizure disorder/history of seizure disorder and/or severe head trauma (other than a single childhood febrile seizure)
* Presence of depression, except for mild depression with no acute episodes and stable condition, as determined by the Investigator
* History of untreated thyroid dysfunction that may be independently associated with cognitive impairment
* Central nervous system-related exclusions:

  1. any medical condition that (per investigator's judgement) would affect subject safety and scientific integrity of the study, e.g., untreated hypothyroidism (TSH >10 mIU/L) or vitamin B12 deficiency (<300 pg/mL) which may contribute to cognitive impairment, delirium, non-AD dementia and other encephalopathies
  2. Hachinski scale score >4 or evidence of stroke within the past 5 years
* Systemic related exclusions:

  1. Active cancer (except squamous cell and basal skin cancers) requiring chemo- or radiation therapy
  2. Positive test results for HIV, HBV, and HCV (unless quantitative PCR negative for HCV) at Screening
  3. Uncontrolled hypertension with a sustained blood pressure >160/100 mmHg at Screening, check-in (Day -1), and prior to the first study drug administration
  4. Fever (body temperature >101.4°F [38.5°C]), acute upper respiratory, or any other infections at Screening, check-in (Day -1), and prior to the first study drug administration
* Any history of drug hypersensitivity, asthma (with the exception of childhood asthma), urticaria or other severe allergic diathesis
* History of adverse - or hypersensitivity reaction to lithium, aspirin, salicylate, L-proline, or any test article excipient
* Female who is breastfeeding, pregnant according to the pregnancy test at Screening or prior to the first study drug administration, or planning to become pregnant during the study
* Magnetic resonance imaging (MRI)-related exclusion criteria (such as intracranial mass, evidence or other anatomical findings that might affect safety or causes of cognitive impairment as assessed by a qualified neurologist)
* History of drug abuse (barbiturate, amphetamine, benzodiazepine, cocaine, opiates and cannabis) within the last 12 months or a positive urine drug screen at Screening or Day -1
* Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements or positive alcohol test at Screening or Day -1.
* More than moderate current alcohol consumption (subjects will be advised to consume no more than 2 units of alcohol/d and completely abstain from 72 hours prior to any visit.
* Treatment with haloperidol, antipsychotics, monoamine oxidase inhibitors, or neuromuscular blocking agents. An appropriate drug-free period will be required for washout, particularly for any especially long half-life drugs.
* Hyponatremia, defined as serum sodium laboratory value outside the standard reference range
* Suspected of having or at risk for Brugada Syndrome
* Prescribed or OTC use of a salicylate-containing product other than low-dose aspirin for cardioprotection (e.g., aspirin, bismuth sub-salicylate, salicylazosulfapyridine [sulfasalazine]) from 1 week before first dose to 1 week after last dosing; any other prescribed anticoagulant medication
* Consumption of poppy seeds or quinine (tonic water) 48 hours prior to Day 1
* Aspirin/nasal polyposis/asthma syndrome
* Participation in a clinical trial and receipt of an investigational medication within 30 days or 5 half-lives (if known), whichever is greater, prior to the first dose of the current study drug.

Inclusion criteria (Healthy Subjects):

* Non-elderly (≥18 and <65 years) and elderly (≥65 and ≤80 years) male and/or female adult subjects of any gender, race or ethnicity, determined to be generally in good physical health
* Willingness to use contraceptive methods as appropriate

Exclusion criteria (Healthy Subjects)

* Clinically significant abnormalities detected by medical history, physical examination, vital sign measurements, ECG findings, or clinical laboratory findings or any historical or present condition/ treatment that may prevent successful or safe study completion, including substance abuse, kidney disease (estimated glomerular filtration rate [eGFR] <60 mL/minute/1.73 m2) or hyponatremia
* Use of any medication on a chronic basis except an oral contraceptive, with appropriate washout of prescription, OTC, vitamins and herbal supplements
* Female pregnant or planning to be pregnant, or breastfeeding

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Alzamend
Locations (2):
- CenExel iResearch, LLC, Decatur, Georgia, United States
- Altasciences, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no pre-specified comparisons between healthy controls and AD patients.
Groups:
- Multiple Ascending Doses of AL001 - Cohort 1: AD-only participants (no normal healthy subjects) were randomized to receive AL001. When adequate safety data were available, a review was done for all participants to make a dose-escalation or dose and/or regimen modification decision. This was repeated for each cohort.
  A total of 8 cohorts received 5 different dose levels of AL001 in multiple ascending doses under fasted conditions up to tolerability/safety limits.
  Cohort 1 included 6 AD subjects only (7 were randomized because 1 subject voluntarily withdrew before dosing); 6 active AD subjects (as per randomization code) received the following treatment or placebo:
  • Cohort 1: 60% of 450 mg lithium carbonate equivalent of AL001 (1890 mg AL001 daily ×14 days, given as 3 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 2a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 2a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults). Blinded results from Cohort 2a were reviewed by the safety review committee before Cohort 2b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 2a: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 2b: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 2b (6 AD subjects). Blinded results from Cohort 2a were reviewed by the safety review committee before Cohort 2b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 2b: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 3a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 3a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults). Blinded results from Cohort 3a were reviewed by the safety review committee before Cohort 3b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 3a: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 3b: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 3b (6 AD subjects). Blinded results from Cohort 3a were reviewed by the safety review committee before Cohort 3b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 3b: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 4a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 4a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults). Blinded results from Cohort 4a were reviewed by the safety review committee before Cohort 4b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 4a: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 4b: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 4b (6 AD subjects). Blinded results from Cohort 4a were reviewed by the safety review committee before Cohort 4b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 4b: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 5a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 5 was planned to be divided into 2 sub-cohorts: Cohort 5a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 5b (8 AD subjects).
  Per randomization, there were 6 active normal healthy subjects in cohort 5a. Stopping rules were invoked by the Safety Committee due to the pharmacokinetic results of Cohort 5a. The Stopping Rules were not invoked due to any adverse event. The stopping criteria were modest increases in plasma levels of lithium and salicylate above what is reported in the literature as the maximum therapeutic range concentrations.
  • Cohort 5a: 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 5b: Subjects for Cohort 5b (6 AD subjects) were not enrolled because the Safety Committee invoked study stopping rules.
  Per randomization, there were 6 active normal healthy subjects in cohort 5a. Stopping rules were invoked by the Safety Committee due to the pharmacokinetic results of Cohort 5a. The Stopping Rules were not invoked due to any adverse event. The stopping criteria were modest increases in plasma levels of lithium and salicylate above what is reported in the literature as the maximum therapeutic range concentrations.
  • Cohort 5b was not dosed. Subjects would have been dosed at 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Combined Placebo Group: 2 subjects were randomized to receive matching placebo (no active drug) concurrently with each of the 8 treatment cohorts. A total of 16 subjects receiving placebo were combined in 1 group.
Period: Overall Study
Arm/Group | Multiple Ascending Doses of AL001 - Cohort 1 | Multiple Ascending Doses of AL001 - Cohort 2a | Multiple Ascending Doses of AL001 - Cohort 2b | Multiple Ascending Doses of AL001 - Cohort 3a | Multiple Ascending Doses of AL001 - Cohort 3b | Multiple Ascending Doses of AL001 - Cohort 4a | Multiple Ascending Doses of AL001 - Cohort 4b | Multiple Ascending Doses of AL001 - Cohort 5a | Multiple Ascending Doses of AL001 - Cohort 5b | Combined Placebo Group
Started | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 16
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 16
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cohort 1 (AD subject), n=6 randomized to AL001(1 withdrawal before dosing). Cohort 2a (healthy volunteers [HV]): n=6 rand. to AL001. Cohort 2b (AD): n=6 rand. to AL001.
  Cohort 3a (HV): n=6 rand. to AL001. Cohort 3b (AD): n=6 rand. to AL001. Cohort 4a (HV): n=6 rand. to AL001. Cohort 4b (AD): n=6 rand. to AL001. Cohort 5 (HV), n=6 rand. to AL001. Combined Placebo Group, n=16.
Groups:
- Multiple Ascending Doses of AL001- Cohort 1 (1890 mg AL001/d, 630mg TID ×14 Days): AD-only participants (no normal healthy subjects) were randomized to receive AL001. When adequate safety data were available, a review was done for all participants to make a dose-escalation or dose and/or regimen modification decision. This was repeated for each cohort.
  A total of 8 cohorts received 5 different dose levels of AL001 in multiple ascending doses under fasted conditions up to tolerability/safety limits.
  Cohort 1 included 6 AD subjects only (7 were randomized because 1 subject voluntarily withdrew before dosing); 6 active AD subjects (as per randomization code) received the following treatment:
  • Cohort 1: 60% of 450 mg lithium carbonate equivalent of AL001 (1890 mg AL001 daily ×14 days, given as 3 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 2a (3150 mg AL001/d, 1050mg TID × 14 Days): The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 2 was divided into 2 sub-cohorts: Cohort 2a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 2b (6 AD subjects). Blinded results from Cohort 2a were reviewed by the safety review committee before Cohort 2b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 2a: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  AL001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 2b (3150 mg AL001/d, 1050mg TID × 14 Days): The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 2 was divided into 2 sub-cohorts: Cohort 2a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 2b (8 AD subjects). Blinded results from Cohort 2a were reviewed by the safety review committee before Cohort 2b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 2b: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  AL001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 3a (4410 mg AL001/d, 1470mg TID × 14 Days): The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 3 was divided into 2 sub-cohorts: Cohort 3a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 3b (6 AD subjects). Blinded results from Cohort 3a were reviewed by the safety review committee before Cohort 3b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 3a: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 3b (4410 mg AL001/d, 1470mg TID × 14 Days): The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 3 was divided into 2 sub-cohorts: Cohort 3a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 3b (6 AD subjects). Blinded results from Cohort 3a were reviewed by the safety review committee before Cohort 3b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 3b: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 4a (5040 mg AL001/d, 1680mg TID × 14 Days): The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 4 was divided into 2 sub-cohorts: Cohort 4a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 4b (6 AD subjects). Blinded results from Cohort 4a were reviewed by the safety review committee before Cohort 4b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 4a: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 4b (5040 mg AL001/d, 1680mg TID × 14 Days): The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 4 was divided into 2 sub-cohorts: Cohort 4a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 4b (6 AD subjects). Blinded results from Cohort 4a were reviewed by the safety review committee before Cohort 4b was randomized. Per randomization, there were 6 active subjects in each cohort:
  • Cohort 4b: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 5a (6300 mg AL001/d, 2100mg TID × 14 Days): The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 5 was planned to be divided into 2 sub-cohorts: Cohort 5a (6 healthy subjects - 3 non-elderly adults and 3 elderly adults) and Cohort 5b (6 AD subjects).
  Per randomization, there were 6 active normal healthy subjects in cohort 5a. Stopping rules were invoked by the Safety Committee due to the pharmacokinetic results of Cohort 5a. The Stopping Rules were not invoked due to any adverse event. The stopping criteria were modest increases in plasma levels of lithium and salicylate above what is reported in the literature as the maximum therapeutic range concentrations.
  • Cohort 5a: 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Multiple Ascending Doses of AL001 - Cohort 5b (6300 mg AL001/d, 2100mg TID × 14 Days): Subjects for Cohort 5b (6 AD subjects) were not enrolled because the Safety Committee invoked study stopping rules due to the pharmacokinetic results of Cohort 5a. The Stopping Rules were not invoked due to any adverse event. The stopping criteria were modest increases in plasma levels of lithium and salicylate above what is reported in the literature as the maximum therapeutic range concentrations.
  • Cohort 5b was not dosed. Subjects would have been dosed at 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product.
- Total: Total of all reporting groups
Arm/Group | Multiple Ascending Doses of AL001- Cohort 1 (1890 mg AL001/d, 630mg TID ×14 Days) | Multiple Ascending Doses of AL001 - Cohort 2a (3150 mg AL001/d, 1050mg TID × 14 Days) | Multiple Ascending Doses of AL001 - Cohort 2b (3150 mg AL001/d, 1050mg TID × 14 Days) | Multiple Ascending Doses of AL001 - Cohort 3a (4410 mg AL001/d, 1470mg TID × 14 Days) | Multiple Ascending Doses of AL001 - Cohort 3b (4410 mg AL001/d, 1470mg TID × 14 Days) | Multiple Ascending Doses of AL001 - Cohort 4a (5040 mg AL001/d, 1680mg TID × 14 Days) | Multiple Ascending Doses of AL001 - Cohort 4b (5040 mg AL001/d, 1680mg TID × 14 Days) | Multiple Ascending Doses of AL001 - Cohort 5a (6300 mg AL001/d, 2100mg TID × 14 Days) | Multiple Ascending Doses of AL001 - Cohort 5b (6300 mg AL001/d, 2100mg TID × 14 Days) | Combined Placebo Group | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 16 | 65
Age, Customized [Mean (Full Range); unit: years] | 63.1 [56 to 71] | 65.4 [52 to 77] | 65.4 [52 to 77] | 57.5 [24 to 72] | 57.5 [24 to 72] | 58.8 [32 to 74] | 58.8 [32 to 74] | 57.3 [33 to 70] |  | 59.4 [24 to 75] | 60.2 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 5 | 1 | 4 | 2 | 4 | 2 |  | 12 | 34
  Male | 7 | 2 | 1 | 5 | 2 | 4 | 2 | 4 |  | 4 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Black or African American | 6 | 0 | 4 | 2 | 4 | 0 | 5 | 0 |  | 7 | 28
  White | 1 | 6 | 2 | 4 | 2 | 6 | 1 | 6 |  | 9 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
Ratio of Plasma Lithium trough >1.0mEq/L or plasma salicylate peak concentrations >30mg/dL [Number; unit: ratio] | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious AEs, TEAEs That Lead to Premature Discontinuation, Abnormal Laboratory Test Results, Abnormal ECG Readings.
Description: To evaluate the safety and tolerability of AL001 in healthy subjects and patients with adverse event(s), AD, descriptive statistics will be presented by treatment group for each cohort and overall, for the following:
  Proportion of participants with treatment-emergent adverse events (TEAEs)
  * Proportion of participants with serious AEs
  * Proportion of participants with TEAEs that lead to premature discontinuation
  * Proportion of participants with abnormal values for each safety laboratory test (change from baseline)
  * Proportion of participants with abnormal values for each Electrocardiogram (ECG) parameter (change from baseline in standard 12-lead ECG parameters)
  For all analyses, placebo-treated subjects from each Cohort were combined (pooled) to provide a composite placebo group for all comparisons. Adverse event profiles for all treated subjects were benign as were placebo-treated subjects. No further statistical analyses were therefore appropriate.
Time Frame: 42 days with a 14-day treatment period
Population: All subjects in the Randomized Analysis Set who received any dose of the study drug. This analysis set was used for all safety analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 1: AD-only participants (no normal healthy subjects) were randomized to receive AL001. When adequate safety data were available, a review was done for all participants to make a dose-escalation or dose and/or regimen modification decision. This was repeated for each cohort.
  A total of 8 cohorts received 5 different dose levels of AL001 in multiple ascending doses under fasted conditions up to tolerability/safety limits.
  Cohort 1 included 8 AD subjects only (9 were randomized because 1 subject voluntarily withdrew before dosing); 6 active and 2 placebo AD subjects (as per randomization code) received the following treatment or placebo:
  • Cohort 1: 60% of 450 mg lithium carbonate equivalent of AL001 (1890 mg AL001 daily ×14 days, given as 3 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 2a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 2 was divided into 2 sub-cohorts: Cohort 2a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 2b (8 AD subjects). Blinded results from Cohort 2a were reviewed by the safety review committee before Cohort 2b was randomized. Per randomization, there were 6 active and 2 placebo subjects in each cohort:
  • Cohort 2a: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 2b: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 2 was divided into 2 sub-cohorts: Cohort 2a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 2b (8 AD subjects). Blinded results from Cohort 2a were reviewed by the safety review committee before Cohort 2b was randomized. Per randomization, there were 6 active and 2 placebo subjects in each cohort:
  • Cohort 2b: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 3a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 3 was divided into 2 sub-cohorts: Cohort 3a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 3b (8 AD subjects). Blinded results from Cohort 3a were reviewed by the safety review committee before Cohort 3b was randomized. Per randomization, there were 6 active and 2 placebo subjects in each cohort:
  • Cohort 3a: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 3b: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 3 was divided into 2 sub-cohorts: Cohort 3a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 3b (8 AD subjects). Blinded results from Cohort 3a were reviewed by the safety review committee before Cohort 3b was randomized. Per randomization, there were 6 active and 2 placebo subjects in each cohort:
  • Cohort 3b: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 4a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 4 was divided into 2 sub-cohorts: Cohort 4a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 4b (8 AD subjects). Blinded results from Cohort 4a were reviewed by the safety review committee before Cohort 4b was randomized. Per randomization, there were 6 active and 2 placebo subjects in each cohort:
  • Cohort 4a: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 4b: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 4 was divided into 2 sub-cohorts: Cohort 4a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 4b (8 AD subjects). Blinded results from Cohort 4a were reviewed by the safety review committee before Cohort 4b was randomized. Per randomization, there were 6 active and 2 placebo subjects in each cohort:
  • Cohort 4b: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 5a: The data from the previous cohort were deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 5 was planned to be divided into 2 sub-cohorts: Cohort 5a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 5b (8 AD subjects).
  Per randomization, there were 6 active and 2 placebo normal healthy subjects in cohort 5a. Stopping rules were invoked by the Safety Committee due to the pharmacokinetic results of Cohort 5a. The Stopping Rules were not invoked due to any adverse event. The stopping criteria were modest increases in plasma levels of lithium and salicylate above what is reported in the literature as the maximum therapeutic range concentrations.
  • Cohort 5a: 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID).
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 vs. Placebo - Cohort 5b: Subjects for Cohort 5b (8 AD subjects) were not enrolled because the Safety Committee invoked study stopping rules due to the pharmacokinetic results of Cohort 5a. The Stopping Rules were not invoked due to any adverse event. The stopping criteria were modest increases in plasma levels of lithium and salicylate above what is reported in the literature as the maximum therapeutic range concentrations.
  • Cohort 5b was not dosed. Subjects would have been dosed at 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation.
- Multiple Ascending Doses of AL001 - Pooled Placebo Group: This is a Cohort which is a composite of all 16 placebo-treated participants derived from all recruited Cohorts.
  Placebo: matching placebo formulation
Arm/Group | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 1 | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 2a | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 2b | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 3a | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 3b | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 4a | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 4b | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 5a | Multiple Ascending Doses of AL001 vs. Placebo - Cohort 5b | Multiple Ascending Doses of AL001 - Pooled Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 16
Participants
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs that lead to premature discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Abnormal values for safety laboratory tests (change from baseline) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 |  | 0
  abnormal ECG parameters (change from baseline) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  No Adverse Events observed | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 |  | 16

2. Secondary Outcome: Maximum Tolerated Dose of AL001 (Lithium Component) in All Subjects Treated With AL001
Description: To characterize the MTD of AL001 in all subjects treated with AL001:
  • Proportion of subjects in each Cohort with plasma trough measurements of lithium > 1.0 mEq/L. Subjects above these values invoke stopping rules for subsequent cohort enrollment.
Time Frame: 42 days with a 14-day treatment period
Population: All subjects in the Safety Analysis Set who received AL001 and had a trough measurement for lithium.
Measure: Number; unit: Proportion of Subjects
Groups:
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 1: Participants were randomized to receive AL001.
  Cohort 1 included 8 AD subjects. In this cohort, 6 active and 2 placebo AD subjects (as per randomization code) received the following treatment or placebo:
  • Cohort 1: 60% of 450 mg lithium carbonate equivalent of AL001 (1890 mg AL001 daily ×14 days, given as 3 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 2a: Steady State Assessment for Trough Plasma Lithium Concentrations
  • Cohort 2a: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 2b: Steady State Assessment for Trough Plasma Lithium Concentrations
  • Cohort 2b: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 3a: Steady State Assessment for Trough Plasma Lithium Concentrations
  • Cohort 3a: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 3b: Steady State Assessment for Trough Plasma Lithium Concentrations
  • Cohort 3b: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 4a: Steady State Assessment for Trough Plasma Lithium Concentrations
  • Cohort 4a: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 4b: Steady State Assessment for Trough Plasma Lithium Concentrations
  • Cohort 4b: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 5a: The data from the previous cohort had to be deemed safe before the next sequential cohort was enrolled and dosing initiated.
  Cohort 5 was planned to be divided into 2 sub-cohorts: Cohort 5a (8 healthy subjects - 4 non-elderly adults and 4 elderly adults) and Cohort 5b (8 AD subjects).
  Modestly higher than threshold lithium plasma concentrations were observed in Cohort 5a and can be expected to occur in AD subjects. It was decided to not run Cohort 5b.
  • Cohort 5a: 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 5b: Cohort 5b was not dosed, because the Safety Committee invoked study stopping rules that were not due to AEs.
  It was decided to not run Cohort 5b.
Arm/Group | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 1 | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 2a | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 2b | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 3a | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 3b | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 4a | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 4b | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 5a | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 5b | Multiple Ascending Doses of AL001 - Pooled Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 16
Proportion of Subjects | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.167 |  | 0

3. Secondary Outcome: Maximum Tolerated Dose of AL001 (Salicylate Component) in All AL001-treated Subjects
Description: To characterize the MTD of AL001 in all subjects:
  • Proportion of all subjects with plasma maximum concentration (Cmax) measurements for salicylate > 30 mg/dL
Time Frame: 42 days with a 14-day treatment period
Population: All subjects in the Safety Analysis Set who received AL001 and had a Cmax measurement for salicylate.
Measure: Number; unit: Proportion of Subjects
Groups:
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 1: Steady State Assessment for Peak Plasma Salicylate Concentrations.
  No healthy subjects were enrolled in Cohort 1. AD Subjects were randomized to receive AL001.
  Cohort 1 included 8 AD subjects. In this cohort, 6 active and 2 placebo AD subjects (as per randomization code) received the following treatment or placebo:
  • Cohort 1: 60% of 450 mg lithium carbonate equivalent of AL001 (1890 mg AL001 daily ×14 days, given as 3 × 210 mg AL001 capsules TID)
  AL 001: a crystal engineered lithium-salicylate-proline lithium delivery product
  Placebo: matching placebo formulation
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 2a: Steady State Assessment for Peak Plasma Salicylate Concentrations
  • Cohort 2a: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 2b: Steady State Assessment for Peak Plasma Salicylate Concentrations
  • Cohort 2b: 100% 450 mg lithium carbonate equivalent of AL001 (3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID).
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 3a: Steady State Assessment for Peak Plasma Salicylate Concentrations
  • Cohort 3a: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 3b: Steady State Assessment for Peak Plasma Salicylate Concentrations
  • Cohort 3b: 140% of 450 mg lithium carbonate equivalent of AL001 (4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 4a: Steady State Assessment for Peak Plasma Salicylate Concentrations
  • Cohort 4a: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in AD Subjects - Cohort 4b: Steady State Assessment for Peak Plasma Salicylate Concentrations
  • Cohort 4b: 160% of 450 mg lithium carbonate equivalent of AL001 (5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID)
- Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 5a: Steady State Assessment for Peak Plasma Salicylate Concentrations.
  Based on the data from Cohort 5a suggested the previous cohort must be deemed safe before the next sequential cohort may be enrolled and dosing initiated.
  It was decided by the safety committee based on stopping rules to not run Cohort 5b.
  • Cohort 5a: 200% of 450 mg lithium carbonate equivalent of AL001 (6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID)
Arm/Group | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 1 | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 2a | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 2b | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 3a | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 3b | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 4a | Multiple Ascending Doses of AL001 in AD Subjects - Cohort 4b | Multiple Ascending Doses of AL001 in Healthy Subjects - Cohort 5a | Multiple Ascending Doses of AL001 - Pooled Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Proportion of Subjects | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.167 | 0

ADVERSE EVENTS:
Time Frame: 42 days with a 14 day treatment period per cohort (phone call follow-up on day 42 to confirm safety)
Groups:
- AD in Cohort 1: Subject w/AD randomized to 1890 mg AL001 daily ×14 days, given as 3 × 210 mg AL001 capsules TID.
- AD on Cohort 2: Subject w/AD randomized to 3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID.
- AD in Cohort 3: Subject w/AD randomized to 4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID.
- AD in Cohort 4: Subject w/AD randomized to 5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID.
- Healthy Subjects in Cohort 2: Healthy Subject randomized to 3150 mg AL001 daily × 14 days, given as 5 × 210 mg AL001 capsules TID.
- Healthy Subjects in Cohort 3: Healthy Subject randomized to 4410 mg AL001 daily × 14 days, given as 7 × 210 mg AL001 capsules TID.
- Healthy Subjects in Cohort 4: Healthy Subject randomized to 5040 mg AL001 daily × 14 days, given as 8 × 210 mg AL001 capsules TID.
- Healthy Subjects in Cohort 5: Healthy Subject randomized to 6300 mg AL001 daily × 14 days - lithium dose equivalent to that used for bipolar/affective disorders, given as 10 × 210 mg AL001 capsules TID.
- AD Subjects on Placebo: Subjects w/AD randomized to Placebo across all Cohorts
- Healthy Subjects on Placebo: Healthy Subjects randomized to Placebo in all Cohorts
Arm/Group | AD in Cohort 1 | AD on Cohort 2 | AD in Cohort 3 | AD in Cohort 4 | Healthy Subjects in Cohort 2 | Healthy Subjects in Cohort 3 | Healthy Subjects in Cohort 4 | Healthy Subjects in Cohort 5 | AD Subjects on Placebo | Healthy Subjects on Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 5/6 | 5/6 | 3/6 | 5/6 | 3/6 | 5/6 | 4/8 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AD in Cohort 1 (N=6) | AD on Cohort 2 (N=6) | AD in Cohort 3 (N=6) | AD in Cohort 4 (N=6) | Healthy Subjects in Cohort 2 (N=6) | Healthy Subjects in Cohort 3 (N=6) | Healthy Subjects in Cohort 4 (N=6) | Healthy Subjects in Cohort 5 (N=6) | AD Subjects on Placebo (N=8) | Healthy Subjects on Placebo (N=8)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (4) | 4 (7) | 2 (5) | 4 (11) | 0 (0) | 3 (8) — Constipation, Abdominal discomfort/distention/pain, nausea, dyspepsia.
Nervous System (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (3) | 2 (4) | 1 (1) | 1 (1) — Headache
Investigations (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) — Hepatic enzyme increased
Renal and Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Pollakisuria
Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (3) — Hypopigmentation, Erythema
Procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Procedural dizziness
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) — Rhinorrhea
Psychiatric (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Insomnia
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Myalgia
Ear Labyrinth (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Tinnitus
Endocrine (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hypothyroidism

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT05363293/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT05363293/SAP_003.pdf